CLINICAL TRIAL: NCT02206308
Title: A Phase I Dose Escalation Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SCT400, a Recombinant Chimeric Anti-CD20 Monoclonal Antibody，in Patients With CD20+ B-cell Non Hodgkin's Lymphoma.
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics of Recombinant Chimeric Anti-CD20 Monoclonal Antibody in Patients With B-cell Non-Hodgkin's Lymphoma.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCT400NHLI
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2013-12

CONDITIONS: B-cell Non Hodgkin's Lymphoma
Keywords: Chimeric anti-CD20 monoclonal antibody(SCT400); escalating doses; safety; pharmacokinetics and pharmacodynamics
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm (Experimental): Three escalating single-dose groups of chimeric anti-CD20 monoclonal antibody(SCT400) : 250 mg/m2 , 375 mg/m2，500 mg/m2, once a week for 4 doses;
  Interventions: Biological: Chimeric anti-CD20 monoclonal antibody

INTERVENTIONS:
Biological: Chimeric anti-CD20 monoclonal antibody
  Other Names: SCT400

SUMMARY:
The purpose of this study is to determine whether SCT400 is safe and effective in the treatment of B-cell Non Hodgkin's lymphoma

ELIGIBILITY:
Inclusion Criteria:

* aged from 18 to 75 years
* having histologically confirmed NHL expressing CD20 antigen
* having relapsed non-Hodgkin's lymphoma(NHL) after at least one prior course of standard therapy
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 according to WHO scale, and expected survival of at least ≥ 3 months
* signed an informed consent form which was approved by the institutional review board of the respective medical center

Exclusion Criteria:

* single measurable lesion ≥7 cm in diameter
* with serious hematologic dysfunction (white blood cell count of <3.0×103/μL; absolute neutrophil count of <1.5×103/ μL; platelet count of < 75×103/μL; hemoglobin level of < 8.0 g/dL; serum immunoglobulin G(IgG) level of <600 mg/dL);, hepatic dysfunction (total bilirubin level of > 1.5×upper limit of normal（ULN）; aspartate amino transferase (AST) and alanine amino transferase (ALT) levels of >2.5 × ULN (≥5 × ULN for patients with liver metastases)); and renal dysfunction (serum creatinine level of > 1.5×ULN )
* having to be at least 4 weeks beyond prior anticancer therapy including corticosteroid, or participating in other clinical trial or have not recovered from significant toxicities of prior therapy
* had received rituximab or other anti-CD20(+) monoclonal antibody treatment within 1 year before enrollment
* had received hematopoietic cytokines, e.g CSF、EPO within 1 week prior to study entry
* with other malignancies ; or central nervous system (CNS) lymphoma, AIDS- related lymphoma; or active opportunistic infection, a serious nonmalignant disease
* having hepatitis B virus surface antigen and /or antibodies to hepatitis C virus or human immunodeficiency virus
* with pleural effusions or ascites secondary to lymphoma; or high risk of tumor lysis syndrome; or recent major surgery (within 28 days )
* with a history of allergic reaction or protein product allergy including murine proteins
* pregnant or lactating or not accepted birth control methods including male patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with infusion-related reaction and with drug-related adverse events. | up to 27 weeks

SECONDARY OUTCOMES:
Area Under the plasma concentration versus time curve (AUC) of SCT400 | prior to the initial dose on day 1 and 0,2,4,8,24,48,72,96,120 hours post-dose

OTHER OUTCOMES:
Time to disease progression | up to 27 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yuan kai Shi, PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Beijing， China